CLINICAL TRIAL: NCT01156233
Title: Endotracheal Tube Tip Position in Orally Intubated 0-4 Year Old Children: Comparative Assessment of the Precision of Two Clinical Techniques
Brief Title: Tube Tip Position in Orally Intubated 0-4year Old Children: Assessment of the Precision of Two Clinical Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Franz Frei (Other)
Responsible Party: Sponsor-Investigator, Franz Frei, Prof. Dr. Franz Frei, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UKBB_ANA_ TET
Record Dates: First submitted 2010-06-30; First posted 2010-07-02 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Intubation, Endotracheal
Keywords: evaluating precision of tube tip position with two methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cuff palpation technique (Experimental): Cuff palpation by the investigator's finger.
  Interventions: Procedure: Anesthesia induction
- Withdrawing tube technique (Experimental): Identification of the tube by withdrawing until good quality breath sounds
  Interventions: Procedure: Anesthesia induction

INTERVENTIONS:
Procedure: Anesthesia induction — Cuff palpation technique: identification of the cuff position in the trachea by palpation.
  Other Names: Pediatric endotracheal tube. Microcuff, Kimberly-Clark.
  Arms: Cuff palpation technique
Procedure: Anesthesia induction — Right mainstem intubation, identification of the tube tip position in the trachea by withdrawing the tube from the right mainstem until good quality breath sound in the left axilla are available.
  Other Names: Pediatric endotracheal tube, Microcuff, Kimberly-Clark
  Arms: Withdrawing tube technique

SUMMARY:
In pediatric anesthesia it is very important to place the endotracheal tube into the right position. This study compares two clinical location methods. The hypothesis means that the two techniques have the same precision of the location of the tip position of a cuffed MICROCUFF (Kimberly-Clark)endotracheal tube.

DETAILED DESCRIPTION:
Appropriate location of the tip of an endotracheal tube (TET), in relation to the carina and vocal cords, is of great importance in pediatric anesthesia. A not optimal laying tube causes life threatening consequences. Therefore, it is very essential to have reliable methods how to place the tube tip in regard of the precision of the localisation. There are no standardized methods how to accomplish a precise position. The study compares two most applied techniques. The first one is the cuff palpation technique (CPT), the second one the deliberate right mainstem intubation technique (RMT).

ELIGIBILITY:
Inclusion Criteria:

* Age 0-4 years
* ASA I-II
* requiring endotracheal tube for surgical/diagnostic procedures

Exclusion Criteria:

* patients with abnormal airway anatomy
* kyphoscoliosis
* syndromes known to affect airway anatomy

Ages: 1 Day to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2010-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Localisation and precision of the tip of the endotracheal tube (TET) in the trachea | 10 minutes
  The study intends to determine the location and precision of the TET within the trachea that results from the use of two techniques. The measurements take place after the induction of the anesthesia and before surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Franz Frei, Professor, Principal Investigator — University Childrens Hospital beider Basel Postfach CH 4005 Basel
Locations (1):
- Universitätskinderspital beider Basel, Basel, Basel, Switzerland